CLINICAL TRIAL: NCT07163884
Title: Adheziv kapsülit tanılı Hastalarda Fasyal Tedavinin ağrı, Normal Eklem Hareket açıklığı, Propriosepsiyon ve Fasya Mimarisine Etkisinin araştırılması
Brief Title: The Effect of Fascial Treatment in Patients With Adhesive Capsulitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Tuğba GÖNEN, Asisst. Prof. Dr., Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025/111
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Adhesive Capsulitis; Ultrasonography; Fascia; Treatment (ProudMe)
Keywords: adhezsiv capsulitis; pain; range of motion; proprioception; fascia architecture
MeSH Terms: conditions — Bursitis; Pain

STUDY DESIGN:
Intervention Model Description: Participants were divided into two groups. Two different interventions were administered to each group. One group will receive electrotherapy and fascia therapy. The other group will receive electrotherapy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascial therapy group (Experimental): In addition to electrotherapy, the patients in the study group will receive a total of five sessions (one day per week for five weeks) of fascial therapy. The protocol will be developed by us. Fascial mobilization will be performed by a trained physiotherapist on the pectoral fascia, deltoid fascia, axillary fascia, and supscapularis fascia, once a week, for 180 seconds each repetition. These sessions will be performed at the pain threshold, and care will be taken to ensure that the pain does not exceed a VAS score of 2.
  Interventions: Other: Facsial therapy
- Control group (Active Comparator): Patients will receive 15 sessions of electrotherapy. A 15-minute hotpack will be applied, followed by a 20-minute TENS application, and then a 6-minute deep heating (1.5 Hz ultrasound) will be applied. Pre-treatment assessments will be repeated after treatment.
  Interventions: Other: electrotherapy treatment

INTERVENTIONS:
Other: electrotherapy treatment — Patients in the electrotherapy group will receive 15 sessions of TENS, hotpack, and ultrasound, 45 minutes each, 5 days a week, for 3 weeks. The treatment program is planned for 20 minutes of TENS, 15 minutes of hotpack, and 10 minutes of ultrasound.
  Arms: Control group
Other: Facsial therapy — In addition to electrotherapy, the patients in the study group will receive a total of five sessions (one day per week for five weeks) of fascial therapy. The protocol will be developed by us. Fascial mobilization will be performed by a trained physiotherapist on the pectoral fascia, deltoid fascia, axillary fascia, and supscapularis fascia, once a week, for 180 seconds each repetition. These sessions will be performed at the pain threshold, and care will be taken to ensure that the pain does not exceed a VAS score of 2.
  Arms: Fascial therapy group

SUMMARY:
Our study is unique in that it utilizes a self-designed fascial mobilization protocol and ultrasonographic evaluation for adhesive capsulitis. Therefore, the aim of our study is to investigate the effects of fascial therapy on pain, normal joint range of motion, proprioception, and fascial architecture in patients diagnosed with adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis (AC) is a common shoulder condition characterized by a gradual increase in spontaneous pain and a limitation in glenohumeral joint range of motion. Its pathophysiology, a pathological process of capsular fibrosis following synovial inflammation, is relatively well understood, but its cause remains unknown. The literature on the treatment of frozen shoulder, whose etiology remains unknown, provides evidence of the effectiveness of conservative treatment approaches such as physiotherapy, analgesics, and steroid injections (1). Pain with movement is minimal in Stage 1 of primary frozen shoulder, while night pain accompanied by activity pain is observed in Stages 2 and 3. Similar pain is observed in secondary frozen shoulder, and the pain is primarily caused by inflammation in the shoulder joint capsule. Increasing range of motion without suppressing pain in patients with frozen shoulder is quite challenging. While heat or electrotherapy are theoretically considered to have positive effects on pain in their treatment, it is difficult to determine the impact of a single method on the natural course of the disease. Therefore, therapeutic methods are generally applied in addition to manual therapy and therapeutic exercises. (2) Pain with movement is minimal in Stage 1 of primary frozen shoulder, while night pain accompanying activity pain is observed in Stages 2 and 3. Similar pain is observed in secondary frozen shoulder, and the pain is primarily caused by inflammation in the shoulder joint capsule. Increasing range of motion without suppressing pain is quite difficult in patients with frozen shoulder. While heat or electrotherapy are considered to have theoretically positive effects on pain in treatment, it is difficult to determine the effect of a single method on the natural course of the disease. Therefore, therapeutic methods are generally applied in addition to manual therapy and therapeutic exercises (3). Studies have suggested the effectiveness of these treatment methods, but sufficient data on the effectiveness of these methods are not yet available (4). Manual therapy methods have begun to be used in adhesive capsulitis, but a meta-analysis has not yet determined the optimal treatment dose (5). Fascia therapy has recently become increasingly used, particularly for lumbar spine pathologies. However, no studies were found on shoulder fascia (6). Ultrasonography is a diagnostic method used in patients with adhesive capsulitis. Ultrasonographic evaluation studies have observed increased coracohumeral ligament thickness, increased supraspinatus tendon thickness, and effusion. However, no ultrasonographic study demonstrating changes in shoulder architecture following physiotherapy interventions was found (7,8). No studies were found on fascial treatment; only one study used instrument-assisted soft tissue mobilization (9). Our study is unique in that it utilized a self-designed fascial mobilization protocol and was evaluated with ultrasonography in adhesive capsulitis. Therefore, the aim of our study was to investigate the effects of fascial treatment on pain, normal joint range of motion, proprioception, and fascial architecture in patients with adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with adhesive capsulitis by a specialist,
* Patients between the ages of 35 and 60,
* Those not diagnosed with cervical disc herniation that could cause other shoulder pathologies,
* Those who have not participated in an upper extremity-related physiotherapy program within the last 6 months,
* Individuals who volunteer to participate in the study,

Exclusion Criteria:

* Individuals who have undergone shoulder surgery consistent with any pathology,
* Individuals with a neurological history,
* Individuals diagnosed with diabetes mellitus (DM)

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Ultrasonographic Measurement | through of the study, average 3 weeks
  An ultrasound (measured by 7.5-10 MHz mobile ultrasound (ALEXUS A10HRL) device will be used to evaluate fascial architecture. The thickness and density of the coracohumeral ligament, supraspinatus tendon, infraspinatus tendon, long head of the biceps, and deltoid fascia, which constitute the patients' shoulder and fascial architecture and are among the structures most affected by adhesive capsulitis, will be evaluated.
The pain | through of the study, average 3 weeks
  Mc Gill Short Form will used to determine the type and severity of the pain. A short form of the McGill Pain Questionnaire (SF-MPQ) has been developed. The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe.
Range of Motion | through of the study, average 3 weeks
  A Universal Goniometer will be used to assess normal range of motion. Measurements will be made regarding shoulder flexion, extension, abduction, adduction, internal and external rotation ranges of motion in three planes of the upper extremity shoulder joint, and the results will be recorded in degrees.
Proprioception | through of the study, average 3 weeks
  Individuals shoulder proprioception will be measured with a laser pointer. A laser pointer is attached to the patient's arm, and the shoulder is flexed 90 degrees, and the laser reflection is marked on the wall. The patient is then asked to close their eyes and maintain the same degree of flexion. The laser reflection is marked. The distance between the two distances is recorded in centimeters. A greater deviation between the two distances indicates a greater loss of proprioception.

SECONDARY OUTCOMES:
Upper extremity functionality | through of the study, average 3 weeks
  The Questionnaire for Arm, Shoulder, and Hand Disabilities (Q-DASH) will be used to assess individuals' upper extremity functions. This questionnaire is a self-administered measurement tool with validated validity and reliability in Turkish. The validity and reliability of the Turkish version of the DASH questionnaire (DASH-T) was conducted in Turkey by Düger et al. in 2006. The questionnaire, consisting of 30 questions, assesses the individual's ability to perform functional activities (21 items), pain (5 items), and psychosocial aspects of the disease (4 items). The total score ranges from 0 to 100, with a higher score indicating better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ager AL, Roy JS, Roos M, Belley AF, Cools A, Hebert LJ. Shoulder proprioception: How is it measured and is it reliable? A systematic review. J Hand Ther. 2017 Apr-Jun;30(2):221-231. doi: 10.1016/j.jht.2017.05.003. PMID 28641738
- [Background] Yakut Y, Yakut E, Bayar K, Uygur F. Reliability and validity of the Turkish version short-form McGill pain questionnaire in patients with rheumatoid arthritis. Clin Rheumatol. 2007 Jul;26(7):1083-7. doi: 10.1007/s10067-006-0452-6. Epub 2006 Nov 15. PMID 17106618
- [Background] Aggarwal A, Saxena K, Palekar TJ, Rathi M. Instrument assisted soft tissue mobilization in adhesive capsulitis: A randomized clinical trial. J Bodyw Mov Ther. 2021 Apr;26:435-442. doi: 10.1016/j.jbmt.2020.12.039. Epub 2020 Dec 31. PMID 33992280
- [Background] Do JG, Hwang JT, Yoon KJ, Lee YT. Correlation of Ultrasound Findings With Clinical Stages and Impairment in Adhesive Capsulitis of the Shoulder. Orthop J Sports Med. 2021 May 10;9(5):23259671211003675. doi: 10.1177/23259671211003675. eCollection 2021 May. PMID 33997079
- [Background] Al Khayyat SG, Falsetti P, Conticini E, Frediani B, Galletti S, Stella SM. Adhesive capsulitis and ultrasound diagnosis, an inseparable pair: a novel review. J Ultrasound. 2023 Jun;26(2):369-384. doi: 10.1007/s40477-022-00725-9. Epub 2022 Oct 25. PMID 36284048
- [Background] Wong KK, Chai HM, Chen YJ, Wang CL, Shau YW, Wang SF. Mechanical deformation of posterior thoracolumbar fascia after myofascial release in healthy men: A study of dynamic ultrasound imaging. Musculoskelet Sci Pract. 2017 Feb;27:124-130. doi: 10.1016/j.math.2016.10.011. Epub 2016 Oct 25. PMID 27847243
- [Background] Kirker K, O'Connell M, Bradley L, Torres-Panchame RE, Masaracchio M. Manual therapy and exercise for adhesive capsulitis: a systematic review with meta-analysis. J Man Manip Ther. 2023 Oct;31(5):311-327. doi: 10.1080/10669817.2023.2180702. Epub 2023 Mar 2. PMID 36861780
- [Background] Nakandala P, Nanayakkara I, Wadugodapitiya S, Gawarammana I. The efficacy of physiotherapy interventions in the treatment of adhesive capsulitis: A systematic review. J Back Musculoskelet Rehabil. 2021;34(2):195-205. doi: 10.3233/BMR-200186. PMID 33185587
- [Background] Kelley MJ, Shaffer MA, Kuhn JE, Michener LA, Seitz AL, Uhl TL, Godges JJ, McClure PW. Shoulder pain and mobility deficits: adhesive capsulitis. J Orthop Sports Phys Ther. 2013 May;43(5):A1-31. doi: 10.2519/jospt.2013.0302. Epub 2013 Apr 30. No abstract available. PMID 23636125
- [Background] Kelley MJ, McClure PW, Leggin BG. Frozen shoulder: evidence and a proposed model guiding rehabilitation. J Orthop Sports Phys Ther. 2009 Feb;39(2):135-48. doi: 10.2519/jospt.2009.2916. PMID 19194024
- [Background] Hsu JE, Anakwenze OA, Warrender WJ, Abboud JA. Current review of adhesive capsulitis. J Shoulder Elbow Surg. 2011 Apr;20(3):502-14. doi: 10.1016/j.jse.2010.08.023. Epub 2010 Dec 16. No abstract available. PMID 21167743